CLINICAL TRIAL: NCT05945992
Title: How to Optimally Train Emotional and Social Skills
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Dr. Sarah Tran-Huu, Principal Investigator, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: TESKx16
Record Dates: First submitted 2023-06-25; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Mental Health
Keywords: Social-emotional learning; Psychological well-being; Subjective well-being; Prevention; Factorial trial
MeSH Terms: conditions — Psychological Well-Being | interventions — Mindfulness; Population Groups

STUDY DESIGN:
Intervention Model Description: Every intervention of each arm will have four components, in varying combination. For each intervention component (mindfulness, self-acceptance, resource activation, emotion regulation) there will exist a control component, when this specific component is not included in the arm.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Condition 1: emotions, self, mindfulness, resources (Experimental): (1) emotion regulation, (2) self-acceptance, (3) mindfulness, (4) resource activation
  Interventions: Behavioral: Emotion regulation; Behavioral: Self-acceptance; Behavioral: Mindfulness; Behavioral: Resource activation
- Condition 2: emotions, self, mindfulness, conflict resolution (Experimental): (1) emotion regulation, (2) self-acceptance, (3) mindfulness, (4) constructive conflict resolution
  Interventions: Behavioral: Emotion regulation; Behavioral: Self-acceptance; Behavioral: Mindfulness; Behavioral: Control component 4_constructive conflict resolution
- Condition 3: emotions, self, stress, resources (Experimental): (1) emotion regulation, (2) self-acceptance, (3) stress management, (4) resource activation
  Interventions: Behavioral: Emotion regulation; Behavioral: Self-acceptance; Behavioral: Resource activation; Behavioral: Control component 3_stress management
- Condition 4: emotions, self, stress, conflict resolution (Experimental): (1) emotion regulation, (2) self-acceptance, (3) stress management, (4) constructive conflict resolution
  Interventions: Behavioral: Emotion regulation; Behavioral: Self-acceptance; Behavioral: Control component 3_stress management; Behavioral: Control component 4_constructive conflict resolution
- Condition 5: emotions, communication, mindfulness, resources (Experimental): (1) emotion regulation, (2) communication skills, (3) mindfulness, (4) resource activation
  Interventions: Behavioral: Emotion regulation; Behavioral: Mindfulness; Behavioral: Resource activation; Behavioral: Control component 2_communication skills
- Condition 6: emotions, communication, mindfulness, conflict resolution (Experimental): (1) emotion regulation, (2) communication skills, (3) mindfulness, (4) constructive conflict resolution
  Interventions: Behavioral: Emotion regulation; Behavioral: Mindfulness; Behavioral: Control component 2_communication skills; Behavioral: Control component 4_constructive conflict resolution
- Condition 7: emotions, communication, stress, resources (Experimental): (1) emotion regulation, (2) communication skills, (3) stress management, (4) resource activation
  Interventions: Behavioral: Emotion regulation; Behavioral: Resource activation; Behavioral: Control component 2_communication skills; Behavioral: Control component 3_stress management
- Condition 8: emotions, communication, stress, conflict resolution (Experimental): (1) emotion regulation, (2) communication skills, (3) stress management, (4) constructive conflict resolution
  Interventions: Behavioral: Emotion regulation; Behavioral: Control component 2_communication skills; Behavioral: Control component 3_stress management; Behavioral: Control component 4_constructive conflict resolution
- Condition 9: group dynamics, self, mindfulness, resources (Experimental): (1) social behavior in groups, (2), self-acceptance, (3) mindfulness, (4) resource activation
  Interventions: Behavioral: Self-acceptance; Behavioral: Mindfulness; Behavioral: Resource activation; Behavioral: Control component 1_social behaviors in groups
- Condition 10: group dynamics, self, mindfulness, conflict resolution (Experimental): (1) social behavior in groups, (2) self-acceptance, (3) mindfulness, (4) constructive conflict resolution
  Interventions: Behavioral: Self-acceptance; Behavioral: Mindfulness; Behavioral: Control component 1_social behaviors in groups; Behavioral: Control component 4_constructive conflict resolution
- Condition 11: group dynamics, self, stress, resources (Experimental): (1) social behavior in groups, (2) self-acceptance, (3) stress management, (4) resource activation
  Interventions: Behavioral: Self-acceptance; Behavioral: Resource activation; Behavioral: Control component 1_social behaviors in groups; Behavioral: Control component 3_stress management
- Condition 12: group dynamics, self, stress, conflict resolution (Experimental): (1) social behavior in groups, (2) self-acceptance, (3) stress management, (4) constructive conflict resolution
  Interventions: Behavioral: Self-acceptance; Behavioral: Control component 1_social behaviors in groups; Behavioral: Control component 3_stress management; Behavioral: Control component 4_constructive conflict resolution
- Condition 13: group dynamics, communication, mindfulness, resources (Experimental): (1) social behavior in groups, (2) communication skills, (3) mindfulness, (4) resource activation
  Interventions: Behavioral: Mindfulness; Behavioral: Resource activation; Behavioral: Control component 1_social behaviors in groups; Behavioral: Control component 2_communication skills
- Condition 14: group dynamics, communication, mindfulness, conflict resolution (Experimental): (1) social behavior in groups, (2) communication skills, (3) mindfulness, (4) constructive conflict resolution
  Interventions: Behavioral: Mindfulness; Behavioral: Control component 1_social behaviors in groups; Behavioral: Control component 2_communication skills; Behavioral: Control component 4_constructive conflict resolution
- Condition 15: group dynamics, communication, stress, resources (Experimental): (1) social behavior in groups, (2) communication skills, (3) stress management, (4) resource activation
  Interventions: Behavioral: Resource activation; Behavioral: Control component 1_social behaviors in groups; Behavioral: Control component 2_communication skills; Behavioral: Control component 3_stress management
- Condition 16: group dynamics, communication, stress, conflict resolution (Active Comparator): (1) social behavior in groups, (2) communication skills, (3) stress management, (4) constructive conflict resolution
  Interventions: Behavioral: Control component 1_social behaviors in groups; Behavioral: Control component 2_communication skills; Behavioral: Control component 3_stress management; Behavioral: Control component 4_constructive conflict resolution

INTERVENTIONS:
Behavioral: Emotion regulation — Psycho-education elements concerning the emergence and functions of emotions, progressive muscle relaxation (PMR), analysis of emotional situations and group exercises
  Arms: Condition 1: emotions, self, mindfulness, resources; Condition 2: emotions, self, mindfulness, conflict resolution; Condition 3: emotions, self, stress, resources; Condition 4: emotions, self, stress, conflict resolution; Condition 5: emotions, communication, mindfulness, resources; Condition 6: emotions, communication, mindfulness, conflict resolution; Condition 7: emotions, communication, stress, resources; Condition 8: emotions, communication, stress, conflict resolution
Behavioral: Self-acceptance — Exercises and guided self-experience targeting heightened knowledge about oneself and acceptance of all personal strengths and weaknesses, exercises based on the internal family systems by R. Schwartz.
  Arms: Condition 10: group dynamics, self, mindfulness, conflict resolution; Condition 11: group dynamics, self, stress, resources; Condition 12: group dynamics, self, stress, conflict resolution; Condition 1: emotions, self, mindfulness, resources; Condition 2: emotions, self, mindfulness, conflict resolution; Condition 3: emotions, self, stress, resources; Condition 4: emotions, self, stress, conflict resolution; Condition 9: group dynamics, self, mindfulness, resources
Behavioral: Mindfulness — Guided mindfulness-exercises, different meditation techniques like body scan, breathing meditation. Reflection and exchange within the group
  Arms: Condition 10: group dynamics, self, mindfulness, conflict resolution; Condition 13: group dynamics, communication, mindfulness, resources; Condition 14: group dynamics, communication, mindfulness, conflict resolution; Condition 1: emotions, self, mindfulness, resources; Condition 2: emotions, self, mindfulness, conflict resolution; Condition 5: emotions, communication, mindfulness, resources; Condition 6: emotions, communication, mindfulness, conflict resolution; Condition 9: group dynamics, self, mindfulness, resources
Behavioral: Resource activation — Exercises focusing on developing positive emotions and fostering personal strengths, based on the Positive Psychology movement of Martin Seligman, working on individual values, life goals and sense of life.
  Arms: Condition 11: group dynamics, self, stress, resources; Condition 13: group dynamics, communication, mindfulness, resources; Condition 15: group dynamics, communication, stress, resources; Condition 1: emotions, self, mindfulness, resources; Condition 3: emotions, self, stress, resources; Condition 5: emotions, communication, mindfulness, resources; Condition 7: emotions, communication, stress, resources; Condition 9: group dynamics, self, mindfulness, resources
Behavioral: Control component 1_social behaviors in groups — Control component for emotion regulation
  Arms: Condition 10: group dynamics, self, mindfulness, conflict resolution; Condition 11: group dynamics, self, stress, resources; Condition 12: group dynamics, self, stress, conflict resolution; Condition 13: group dynamics, communication, mindfulness, resources; Condition 14: group dynamics, communication, mindfulness, conflict resolution; Condition 15: group dynamics, communication, stress, resources; Condition 16: group dynamics, communication, stress, conflict resolution; Condition 9: group dynamics, self, mindfulness, resources
Behavioral: Control component 2_communication skills — Control component for self-acceptance
  Arms: Condition 13: group dynamics, communication, mindfulness, resources; Condition 14: group dynamics, communication, mindfulness, conflict resolution; Condition 15: group dynamics, communication, stress, resources; Condition 16: group dynamics, communication, stress, conflict resolution; Condition 5: emotions, communication, mindfulness, resources; Condition 6: emotions, communication, mindfulness, conflict resolution; Condition 7: emotions, communication, stress, resources; Condition 8: emotions, communication, stress, conflict resolution
Behavioral: Control component 3_stress management — Control component for mindfulness
  Arms: Condition 11: group dynamics, self, stress, resources; Condition 12: group dynamics, self, stress, conflict resolution; Condition 15: group dynamics, communication, stress, resources; Condition 16: group dynamics, communication, stress, conflict resolution; Condition 3: emotions, self, stress, resources; Condition 4: emotions, self, stress, conflict resolution; Condition 7: emotions, communication, stress, resources; Condition 8: emotions, communication, stress, conflict resolution
Behavioral: Control component 4_constructive conflict resolution — Control component for resource activation
  Arms: Condition 10: group dynamics, self, mindfulness, conflict resolution; Condition 12: group dynamics, self, stress, conflict resolution; Condition 14: group dynamics, communication, mindfulness, conflict resolution; Condition 16: group dynamics, communication, stress, conflict resolution; Condition 2: emotions, self, mindfulness, conflict resolution; Condition 4: emotions, self, stress, conflict resolution; Condition 6: emotions, communication, mindfulness, conflict resolution; Condition 8: emotions, communication, stress, conflict resolution

SUMMARY:
The goal of this clinical trial is to compare different well-being intervention components in healthy individuals. The main question it aims to answer is how an optimal emotional and social learning program should be composed. Participants will participate in one of 16 courses over 14-weeks which will have a varying combination of four components:

* emotion regulation,
* mindfulness,
* self-acceptance and
* resource activation.

For each of these components there will be a control component. Further, there will be a waitlist-control-group included.

DETAILED DESCRIPTION:
Background: Social-emotional skills are of great importance for academic and professional success and are a huge protective factor of mental health.

Objectives: The aim of the study therefore is to examine the optimal combination of different well-being intervention components to foster mental health and subjective well-being in a student and trainee population. The investigators draw on current concepts like mindfulness which already proved to be empirically effective and try to compare their effectiveness and understand how they work together, whether they strengthen or complement each other.

Methods: In a factorial design trial with 16 different intervention conditions, up to 240 students or trainees will participate in a 14-week well-being-intervention. This intervention with a maximum of 15 participants per course consists of weekly 1,5h sessions plus 3 full-day appointments using psycho-educational elements, practical exercises and group discussion on various topics. Participants will complete online surveys on subjective and psychological well-being, mental health, and several resilience factors pre-, during and post-intervention as well as 5 months after completion as follow-up assessments.

Implications: The study will contribute to an evidence-based and easily accessible and scalable well-being intervention, supporting health promotion and stress prevention in the general population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Fluent in German language
* Student at a German university or trainee in vocational training

Exclusion Criteria:

* Acute mental health crisis (e.g., suicidality)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in emotional regulation, measured by self-appraisal of emotional skills | baseline (pre), 7-8 weeks (intermediate), 14 weeks (post), 6 months (first follow-up), 9 months (second follow-up)
  27 items in total, 3 items per 9 subscales (attention, body perception, clarity, understanding, regulation, acceptance, resilience, self support, willingness of confrontation) (German instrument: Selbsteinschätzung emotionaler Kompetenzen, SEK-27, Berking & Znoj, 2011)
  Scores range from 0 ("not at all") to 4 ("(almost) always").; higher scores reflect higher assessment of emotional skill.
Change in self-efficacy, measured by scale on general self-efficacy | baseline (pre), 7-8 weeks (intermediate), 14 weeks (post), 6 months (first follow-up), 9 months (second follow-up)
  10 items on one-dimensional scale. (German instrument; Skala zur Allgemeinen Selbstwirksamkeitserwartung, SWE, Jerusalem & Schwarzer, 2003)
  Scores range from 1 ("strongly disagree") to 4 ("strongly agree"); higher scores reflect higher self-efficacy.
Change in psychological well-being, measured by the Psychological Wellbeing Scale (German version) | baseline (pre), 7-8 weeks (intermediate), 14 weeks (post), 6 months (first follow-up), 9 months (second follow-up)
  6 subscales (autonomy, environmental mastery, purpose in life, personal growth, relations with others, self-acceptance) (German Version of the PWB Scale by Ryff et al. 2007; Fragebogen zum Psychologischen Wohlbefinden, Risch, Strohmayer & Stangier, 2005)
  Scores range from 1 ("strongly disagree") to 6 ("strongly agree"); higher scores reflect better well-being.
Change in mindfulness, measured by the Mindfulness Attention and Awareness Scale (German Version) | baseline (pre), 7-8 weeks (intermediate), 14 weeks (post), 6 months (first follow-up), 9 months (second follow-up)
  15 items on one-dimensional scale (Michalak, Heidenreich, Ströhle & Nachtigall, 2011)
  Scores range from 1 ("almost always") to 6 ("almost never") assessing daily exercises and activities; higher scores reflect lower mindfulness.
Change in flourishing, measured by Flourishing Scale (German version) | baseline (pre), 7-8 weeks (intermediate), 14 weeks (post), 6 months (first follow-up), 9 months (second follow-up)
  8 items on one-dimensional scale (Esch et al., 2013)
  Scores range from 1 ("stongly disagree") to 7 ("strongly agree"); higher scores reflect higher appraisal of flourishing in life.
Change in self-compassion, measured by the Self-Compassion Scale (German version) | baseline (pre), 7-8 weeks (intermediate), 14 weeks (post), 6 months (first follow-up), 9 months (second follow-up)
  26 items measuring 6 scales (self-kindness, self-judgment, common humanity, isolation, mindfulness, over-identification) (Hupfeld & Ruffieux, 2011)
  Scores range from 1 ("very seldom") to 5 ("very often") assessing daily exercises and activities; higher scores reflect higher self-compassion.
Change in perceived stress, measured by the Perceived Stress Scale (German version) | baseline (pre), 7-8 weeks (intermediate), 14 weeks (post), 6 months (first follow-up), 9 months (second follow-up)
  10 items; 6 items assessing helplessness, and 4 items assessing self-efficacy. (Schneider et al., 2020)
  Scores range from 1 ("never") to 5 ("very often") ; higher scores reflect higher perceived stress.

SECONDARY OUTCOMES:
Change in subjective well-being, measured by the Positive and Negative Affective Schedule (PANAS) | baseline (pre), 7-8 weeks (intermediate), 14 weeks (post), 6 months (first follow-up), 9 months (second follow-up)
  The scale consists of a total of 20 items, when 10 items referring to positive affect, 10 items referring to negative affect.
  Scores range from 1 ("not at all") to 5 ("extremely") assessing the experience of positive or negative emotional states during the past week; higher scores reflect higher experiencing of this emotion.
Change in subjective life-satisfaction | baseline (pre), 7-8 weeks (intermediate), 14 weeks (post), 6 months (first follow-up), 9 months (second follow-up)
  5 items on one-dimensional scale (Schumacher 2003)
  Scores range from 1 ("not at all") to 7 ("extremely"); higher scores reflect higher life satisfaction.
Change in mental health, measured by the Patient Health Questionnaire (German version, by Löwe, Zipfel & Herzog, 2002) | baseline (pre), 7-8 weeks (intermediate), 14 weeks (post), 6 months (first follow-up), 9 months (second follow-up)
  The sum of the PHQ-9 is used to assess general mental health. Scales concerning 1. somatic symptoms: assessing body symptoms, scores range from "not impaired" to 3 ("strongly impaired") / 2. depression: 9 items, scores from 0 "not at all" to 3 "almost every das / 3. anxiety: items assessing panic attac or other forms of anxiety, scores "Yes" or "No", respectively assessing general nervousness and anxiety from 1 ("not at all") to 3 ("on more than half days in the week"), higher scores meaning higher symptomatology / 4. eating disorder: items assessing eating difficulties and feelings of uncontrollability, (Yes vs. No"). Yes-answers on all items indicating eating disorder / 5. alcohol misuse: items assessing drinking patterns, scores "yes" vs. "no", when at least 1 item is answered with a "yes", misuse ist assessed / 6. psychosocial functionality: 1 item on the impairment of those symptomes, from 1 ("not at all impaired") to 4 ("very highly impaired")

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Wälde, Prof. Dr., Study Chair — Chair in Macroeconomics, JGU Johannes Gutenberg Universität Mainz

IPD SHARING:
Plan to Share IPD: Yes
Anonymized answers to questionnaires (all data)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: as soon as results are available (expected fall 2024)
Access Criteria: on web page once paper is published